CLINICAL TRIAL: NCT01964755
Title: Phase II Study of Chemotherapy (Doxorubicin, Methotrexate and Leucovorin) in Combination With Antiviral-Based Therapy (Zidovudine + Hydroxyurea) for AIDS, Immunocompromised, or Immunocompetent Patients With Relapsed or CNS Positive Epstein Barr Virus Associated Lymphoma
Brief Title: Chemotherapy for Relapsed Epstein Barr Virus Associated Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Investigator Decision
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Juan C. Ramos, Associate Professor of Clinical, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20090166
Record Dates: First submitted 2013-10-14; First posted 2013-10-17 (Estimated); Results first posted 2019-09-23 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-08

CONDITIONS: Epstein Barr Virus Associated Non Hodgkin's Lymphoma; Epstein Barr Virus Associated Hodgkin's Lymphoma; Post-Transplant Lymphoproliferative Disease
Keywords: EBV+; NHL; HL; Non Hodgkin's Lymphoma; Hodgkin's Lymphoma; Epstein Barr Virus; Epstein Barr Virus Associated Non Hodgkin's Lymphoma; Epstein Barr Virus Associated Hodgkin's Lymphoma; Post-Transplant Lymphoproliferative Disease
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Hodgkin Disease; Epstein-Barr Virus Infections | interventions — Doxorubicin; Methotrexate; merphos; Leucovorin; Hydroxyurea; Zidovudine; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Chemotherapy + Antiviral-Based Therapy (Experimental): Combination Chemotherapy for up to six (6) 21-day cycles and Antiviral-Based Therapy:
  * Chemotherapy: Up to 6 cycles, 21 days each:
    * Doxorubicin: 20 mg/m2 intravenously (IV) on Day 1 per study protocol;
    * Rituximab: 375mg/m2 (optional) IV on Day 1 per study protocol;
    * Methotrexate: 3.5 gm/m2 IV on Day 2 per study protocol;
    * Leucovorin: 10 mg/m2 IV starting approximately 24 hours after start of Methotrexate infusion, and then 25 mg orally every 6 hours for at least 10 doses per study protocol;
  * Antiviral-Based Therapy
    * Zidovudine: Starting 750 mg/m2 IV on Day 2, then 1200 mg orally twice daily for 10 doses per study protocol;
    * Hydroxyurea: 1,000 mg orally twice daily starting Day 2 for a total of 10 doses per study protocol.
  Interventions: Drug: Doxorubicin; Drug: Methotrexate; Drug: Leucovorin; Biological: Hydroxyurea; Drug: Zidovudine; Drug: Rituximab

INTERVENTIONS:
Drug: Doxorubicin — Doxorubicin 20 mg/m2 intravenously will be administered on Day 1 in patients with systemic (non-primary CNS) lymphoma as per institutional guidelines
  Other Names: Adriamycin
Drug: Methotrexate — Methotrexate administered starting on Day 2, per study protocol.
  Other Names: Methotrexate sodium; Mexate; Mexate-aq; Folex; Abitrexate; Rheumatrex; Amethopterin
Drug: Leucovorin — Leucovorin administered first intravenously 24 hours after start of Methotrexate infusion, then orally every 6 hours for at least 10 doses, per study protocol.
  Other Names: Leucovorin Calcium; Wellcovorin; Citrovorum Factor; Folinic Acid; 5-formyl tetrahydrofolate; LV; LCV
Biological: Hydroxyurea — Hydroxyurea administered orally twice daily starting on Day 2, and continuing for a total of 10 doses, per study protocol
  Other Names: Hydroxycarbamide (rINN); Hydrea
Drug: Zidovudine — Zidovudine administered first intravenously on Day 2, and then orally twice daily for 10 doses, per study protocol.
  Other Names: Retrovir; Azidothymidine (AZT)
Drug: Rituximab — Rituximab is optional and will be administered to study participants, per study protocol.
  Other Names: Rituxan

SUMMARY:
By combining a variety of agents that potentiate Zidovudine (ZDV), the investigators hope to induce remission in this generally fatal disease. Most therapies for aggressive B cell lymphomas are based upon intensive chemotherapeutic regimens, expensive modalities (bone marrow transplant, Rituximab), or experimental approaches (gene therapy, cytotoxic T cell infusion) that are difficult to implement in heavily pre-treated patients. Therapy for relapsed aggressive B cell lymphomas is very poor. Even curable lymphomas such as Burkitt Lymphoma (BL) and Hodgkin lymphoma are extremely difficult to treat in relapse and/or after stem cell transplant failure. The investigators propose a novel therapeutic approach that exploits the presence of Epstein-Barr virus (EBV) in lymphomas; antiviral mediated suppression of NF-kB and disruption of viral latency.

ELIGIBILITY:
Inclusion Criteria:

1. Any stage, histologically or cytologically documented intermediate to high grade relapsed or refractory EBV+ non-Hodgkin's (NHL) or Hodgkin's lymphoma (HL), or any treated or untreated patients with EBV+ lymphoma involving CNS. Patients with relapsed or refractory monomorphic (monoclonal) post-transplant lymphoproliferative disease (PTLD) are also eligible.
2. Patients who are HIV+ or negative. Documentation of HIV infection can be done at any time prior to study entry. Documentation may be serologic (positive ELISA and positive Western blot), molecular (positive HIV viral RNA), or other federally approved licensed HIV test. Prior documentation of HIV seropositivity is acceptable.
3. Tumors must be positive for EBV. This may be done either by Epstein-Barr virus-encoded small RNA (EBER) stain on the original tumor or the biopsy of relapsed disease (if performed). Biopsy of relapsed disease is desirable but not mandatory. If stains for Epstein-Barr virus latent membrane protein 1 (LMP1) done outside are positive, EBER does not need to be done.
4. All patients, except those who have CNS involvement, must have relapsed or progressed from at least one previous chemotherapy based regimen.
5. Measurable or non-measurable tumor parameter(s). Non-measurable tumor parameter(s) is defined as not having bi-dimensional measurements (e.g., gastric or marrow involvement), but can be followed for response by other diagnostic tests such as gallium scan, Positron emission tomography (PET) imaging and/or bone marrow biopsy.
6. Age ≥ 18 years.
7. Karnofsky performance status (KPS) ≥ 50%/Eastern Cooperative Oncology Group (ECOG) Performance Score 0, 1, 2.
8. Patients must have adequate end organ and bone marrow function as defined below:

   * 8.1 Absolute neutrophil count ≥ 1,500 cells/mm3 and platelets ≥ 75,000 cells/dL unless cytopenias are secondary to lymphomatous involvement of bone marrow or due to HIV-related thrombocytopenia. All patients must be off colony stimulating factor therapy at least 24 hours prior to institution of Cycle 1 chemotherapy.
   * 8.2 Adequate hepatic function: Serum glutamic-oxaloacetic transaminase (SGOT) ≤ 5 times the upper limit of normal. Total bilirubin ≤ 2.0 mg/dL (unless elevated secondary to lymphomatous involvement of liver or biliary system or due to other HIV medications [e.g., indinavir, tenofovir or atazanavir]). Patients who are negative for Hepatitis B, or if infected with Hepatitis B, receiving anti-Hepatitis B therapy are eligible. All subjects will be required to be screened for Hepatitis B and C. Per Infectious Diseases Society of America (IDSA) and American Association for the Study of Liver Diseases (AASD) guidelines, those subjects that show no immunity, defined by the lack of Hepatitis B surface antibody, and show evidence of chronic infection (i.e. HBsAg+, HBcore+, HBsAB-) will be required to be on anti-Hepatitis B therapy, during the study, in order to be eligible. Patients will be permitted to enroll in the study provided liver function tests meet criteria listed above, and there is no evidence of cirrhosis. The exact Hepatitis B therapy will be at the discretion of the infection disease specialist or investigator. However all patients who present with acute hepatitis B or show normal transaminases and are HBsAg+ and IgM+ for Hepatitis core antigen will not be eligible for trial enrollment. Subjects who are Hepatitis C antibody positive, with or without a positive Hepatitis C RNA level, will be permitted to enroll in the study provided liver function tests meet criteria listed above, and have no evidence of cirrhosis. Patients diagnosed with Hepatitis C less than 6 months from trial enrollment, will be considered to have Acute Hepatitis C and will be excluded from study unless Hep C viral load is undetectable.
   * 8.3 Creatinine ≤ 2.0 mg/dL or creatinine clearance ≥ 60 mL/min unless due to renal involvement by lymphoma.
9. Concurrent radiation, with or without steroids, for emergency conditions secondary to lymphoma (CNS tumor, cord compression, etc.) will be permitted.
10. Females with childbearing potential must have a negative serum pregnancy test within 7 days prior of entering into the study. Men and women must agree to use adequate birth control if conception is possible during the study. Women must avoid pregnancy and men avoid fathering children while in the study and for 6 months following the last study drug treatment.
11. Able to give consent.
12. Patients already receiving erythropoietin or Granulocyte-colony stimulating factor (G-CSF) are eligible, although G-CSF therapy must be discontinued at least 24 hours prior to receiving chemotherapy.
13. The maximum cumulative dose of doxorubicin allowed is 450 mg/m2. Patients who have previously received doxorubicin with a cumulative dose of 350 mg/m2 or greater are eligible but MAY NOT receive doxorubicin under protocol.

Exclusion Criteria:

1. Concurrent active malignancies, with the exception of in situ carcinoma of the cervix, non-metastatic, non-melanomatous skin cancer, or Kaposi sarcoma not requiring systemic chemotherapy.
2. Myocardial infarction (MI) within 6 months prior to study entry, New York Heart Association (NYHA) Class II or greater heart failure, uncontrolled angina, severe, uncontrolled ventricular arrhythmias, clinically significant pericardial disease, or electrocardiograph evidence of acute ischemic or active conduction system abnormalities.
3. Left Ventricular Ejection Fraction (LVEF) that is less than the lower institutional limits of normal as assessed by Multiple Gated Acquisition (MUGA) scan or echocardiogram within 6 weeks prior to registration.
4. Subjects with viral hepatitis who do not meet the criteria listed on (8.2) will be not be eligible. All patients who present with acute hepatitis B including those with normal transaminases who are HBsAg+ and IgM + for hepatitis core antigen will not be eligible. Subjects who are Hepatitis B core antibody positive are eligible only if they start or are on prophylactic therapy. A hepatitis B viral load should be confirmed negative on all patients who are hepatitis B core antibody positive, but hepatitis B antigen negative. Patients refusing to take any anti-hepatitis B therapy during study will also be excluded. Patients diagnosed with Hepatitis C are eligible if they meet criteria listed on (8.2).
5. Psychological, familial, sociological or geographical conditions that do not permit treatment and/or medical follow-up required to comply with the study protocol.
6. Patients may not be receiving any other investigational agents.
7. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements. Patients with mycobacterium avium will not be excluded.
8. Pregnant or breast-feeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2009-04-21 (Actual); Primary Completion 2018-06-07 (Actual); Study Completion 2018-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Juan Carlos Ramos, MD, Study Chair — University of Miami
Locations (2):
- United States (2):
  - University of Miami, Miami, Florida
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina

RESULTS

PARTICIPANT FLOW:
Groups:
- Chemotherapy + Antiviral-Based Therapy: Combination Chemotherapy for up to six (6) 21-day cycles and Antiviral-Based Therapy per study protocol:
  * Chemotherapy: Up to 6 cycles, 21 days each:
    * Doxorubicin: 20 mg/m2 intravenously (IV) on Day 1;
    * Rituximab: 375mg/m2 (optional) IV on Day 1;
    * Methotrexate: 3.5 gm/m2 IV on Day 2;
    * Leucovorin: 10 mg/m2 IV starting approximately 24 hours after start of Methotrexate infusion, and then 25 mg orally every 6 hours for at least 10 doses;
  * Antiviral-Based Therapy
    * Zidovudine: Starting 750 mg/m2 IV on Day 2, then 1200 mg orally twice daily for 10 doses;
    * Hydroxyurea: 1,000 mg orally twice daily starting Day 2 for a total of 10 doses.
  Doxorubicin: Doxorubicin 20 mg/m2 intravenously will be administered on Day 1 in patients with systemic (non-primary CNS) lymphoma as per institutional guidelines
  Methotrexate: Methotrexate administered starting on Day 2.
Period: Overall Study
Arm/Group | Chemotherapy + Antiviral-Based Therapy
Started | 6
Cycle 2 | 5
Cycle 3 | 4
Cycle 4 | 4
Cycle 5 | 4
Completed | 4
Not Completed | 2
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Arm/Group | Chemotherapy + Antiviral-Based Therapy
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 1
Age, Continuous [Median (Full Range); unit: years] | 47 [33 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Rate of Complete Response to Protocol Therapy
Description: Complete Response (CR) rate in study participants to protocol therapy. Response will be assessed via CT Scan and bone marrow aspirate/biopsy, if applicable. Complete response criteria include:
  * Complete disappearance of all detectable clinical and radiographic evidence of disease and disappearance of all disease-related symptoms if present before therapy, and normalization of those biochemical abnormalities definitely assignable to Non Hodgkin's Lymphoma (NHL);
  * All lymph nodes and tumor masses disappeared or regressed to normal size (≤ 1.5 cm in their greatest transverse diameters for nodes > 1.5 cm before therapy);
  * Previously involved nodes that were 1.1 to 1.5 cm in their greatest transverse diameter (GTD) before treatment must have decreased to ≤ 1 cm in their GTD after treatment, or by more than 75% bin the sum of the products of the greatest diameters (SPD);
  * No new sites of disease.
Time Frame: About 21 days
Population: Participants who started at least one cycle of protocol therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy + Antiviral-Based Therapy
Number analyzed (Participants) | 6
Participants | 3

2. Secondary Outcome: One-year Rate of Overall Survival
Description: Rate of overall survival of study participants at one year since initiation of protocol therapy. Overall survival (OS) will be measured from the date of initiation of study treatment until date of death from any cause. In the absence of death, the follow-up will be censored at date of last contact (censored observation). Kaplan-Meier estimate of overall survival at one-year.
Time Frame: 12 months
Population: Participants receiving at least one cycle of protocol therapy.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemotherapy + Antiviral-Based Therapy
Number analyzed (Participants) | 6
percentage of participants | 83.3 [27.3 to 97.5]

3. Secondary Outcome: One-Year Rate of Failure-Free Survival (FFS)
Description: Rate of failure-free survival of study participants one-year after start of protocol therapy. Failure-free survival (FFS) will be measured from the date of treatment initiation until date of documented disease progression, relapse after response, or death from any cause. For patients alive and free of relapse or progression, follow-up time will be censored at the last documented date of failure-free status. Kaplan-Meier estimate of failure-free survival at one-year.
Time Frame: 12 months
Population: Participants receiving at least one cycle of protocol therapy.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemotherapy + Antiviral-Based Therapy
Number analyzed (Participants) | 6
percentage of participants | 37.5 [1.1 to 80.8]

4. Secondary Outcome: Rate of Toxicity Related to Protocol Therapy
Description: Rate of adverse events, serious adverse events or other toxicities related to protocol therapy in study participants.
Time Frame: Through Duration of Protocol Therapy, Up to six 21-day cycles (+/- 7 days)
Population: Participants starting at least once cycle of protocol therapy. Participants experiencing toxicity are tabulated by grade (gr.) of toxicity.
Measure: Count of Participants; unit: Participants
Arm/Group | Chemotherapy + Antiviral-Based Therapy
Number analyzed (Participants) | 6
Participants
  Patients w/Toxicity Definitely Treatment-Related | 0
  Gr. 4 Toxicity Probably/Possibly Treatment-Related | 1
  Gr. 3 Toxicity Probably/Possibly Treatment-Related | 4
  Gr. 2 Toxicity Probably/Possibly Treatment-Related | 6
  Gr. 1 Toxicity Probably/Possibly Treatment-Related | 6

5. Secondary Outcome: HIV Viral Load in Positive Subjects Before, During and After Protocol Therapy
Description: Measurement of HIV Viral Load in positive subjects before, during and after protocol therapy to assess the effect of protocol therapy on immune reconstitution or exhaustion.
Time Frame: From Baseline Up to 1 Year Post-Therapy
Population: Per protocol, evaluable participants are those who receive 3 or more cycles of treatment. Three of these participants were HIV-positive. Before therapy, HIV viral load was undetectable in 2 participants.
Measure: Number; unit: copies/ml
Arm/Group | Chemotherapy + Antiviral-Based Therapy
Number analyzed (Participants) | 3
copies/ml
  Before Therapy: number analyzed (Participants) | 1
  Before Therapy | 333
  During Therapy | NA — HIV viral load undetectable in study participants.
  After Therapy | NA — HIV viral load undetectable in study participants.

6. Secondary Outcome: T-Cell Subset Levels in Peripheral Blood in Positive Participants Before, During and After Protocol Therapy
Description: Measurement of T-cell subset levels (CD4, CD8) in peripheral blood before, during and after protocol therapy to assess the effect of protocol therapy on immune re-constitution or exhaustion.
Time Frame: From Baseline Up to 1 Year Post-Therapy
Population: Per protocol, evaluable participants are those who receive 3 or more cycles of treatment. Three of these participants were HIV-positive. Data for T-cell subset levels (CD4, CD8) were available during and after for two of these three participants.
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Chemotherapy + Antiviral-Based Therapy
Number analyzed (Participants) | 3
cells/mm^3
  CD4 count, Before Therapy | 328 (164.05)
  CD4 count, During Therapy: number analyzed (Participants) | 2
  CD4 count, During Therapy | 285 (124.58)
  CD4 count, After Therapy: number analyzed (Participants) | 2
  CD4 count, After Therapy | 323.5 (178.90)
  CD8 count, Before Therapy | 1246 (668.86)
  CD8 count, During Therapy: number analyzed (Participants) | 2
  CD8 count, During Therapy | 1006 (741.05)
  CD8 count, After Thaerapy: number analyzed (Participants) | 2
  CD8 count, After Thaerapy | 1006 (741.05)

7. Secondary Outcome: EBV Viral Load in Peripheral Blood Before, During and After Protocol Therapy
Description: Measurement of Epstein Barr Virus (EBV) viral load in peripheral blood in study participants before, after treatment, and during surveillance in order to correlate the presence of with tumor load and disease status.
Time Frame: From Baseline Up to 1 year Post-Therapy
Population: Serum EBV viral load levels were below the limit of detection in subjects before therapy. Data were not collected during and after therapy.
Arm/Group | Chemotherapy + Antiviral-Based Therapy
Number analyzed (Participants) | 0

8. Secondary Outcome: EBV Reactivation in Circulating Peripheral Blood Memory B-cells Before and After Protocol Therapy.
Description: Measurement of EBV reactivation in circulating peripheral blood memory B-cells before and after treatment with chemotherapy/Zidovudine (ZDV) in order to assess the drug effect on EBV latency.
Time Frame: From Baseline Up to 1 year Post-Therapy
Population: This outcome measure was added via amendment for new participants enrolled after December 2016 however; no new participants were enrolled. No data were collected for this outcome measure.
Arm/Group | Chemotherapy + Antiviral-Based Therapy
Number analyzed (Participants) | 0

9. Secondary Outcome: Baseline Tumor EBV Gene Expression Profile in Study Participants
Description: Determine baseline tumor EBV gene expression profile to assess viral thymidine kinases. (BXLF1/vTK and BGLF4/PK), EBV latency pattern (I, II or III) and lytic phase.
Time Frame: Baseline
Population: as for outcome 8
Arm/Group | Chemotherapy + Antiviral-Based Therapy
Number analyzed (Participants) | 0

10. Secondary Outcome: Measurement of Immune Activation Markers and Inflammation in Peripheral Blood
Description: Measurement of immune activation markers and inflammation in peripheral blood in response to treatment and EBV reactivation.
Time Frame: Through Duration of Response to Protocol Therapy Until Disease Progression, Up to 5 years
Population: as for outcome 8
Arm/Group | Chemotherapy + Antiviral-Based Therapy
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 4 years
Arm/Group | Chemotherapy + Antiviral-Based Therapy
All-Cause Mortality (participants affected / at risk) | 2/6
Serious Adverse Events (participants affected / at risk) | 2/6
Other Adverse Events (participants affected / at risk) | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy + Antiviral-Based Therapy (N=6)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Platelet count decreased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy + Antiviral-Based Therapy (N=6)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Alanine aminotransferase increased (Metabolism and nutrition disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 6 (23)
Anorexia (Metabolism and nutrition disorders) | 3 (4)
Anxiety (Psychiatric disorders) | 1 (1)
Aspartate aminotransferase increased (Metabolism and nutrition disorders) | 2 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (4)
Blood bilirubin increased (Investigations) | 1 (4)
Conjunctivitis infective (Infections and infestations) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Creatinine increased (Investigations) | 2 (6)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (4)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Fatigue (General disorders) | 2 (2)
Fever (General disorders) | 1 (1)
Flushing (Skin and subcutaneous tissue disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (3)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Headache (General disorders) | 2 (4)
Hiccups (Reproductive system and breast disorders) | 3 (6)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 6 (47)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (2)
Hypernatremia (Metabolism and nutrition disorders) | 3 (4)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (9)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (10)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (4)
Hypokalemia (Metabolism and nutrition disorders) | 4 (18)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (3)
Hyponatremia (Metabolism and nutrition disorders) | 3 (6)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Hypoxia (Reproductive system and breast disorders) | 1 (1)
INR increased (Investigations) | 1 (1)
Insomnia (General disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Leukocytes (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Lymphocyte count decreased (Investigations) | 3 (12)
Malaise (General disorders) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 3 (12)
Nausea (Gastrointestinal disorders) | 5 (16)
Neutrophil count decreased (Investigations) | 2 (5)
Oral pain (General disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Personality change (Nervous system disorders) | 1 (1)
Pharyngolaryngeal pain (General disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Seborrheic Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Genital Herpes (Infections and infestations) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (7)
Weight loss (General disorders) | 1 (1)
White blood cell decreased (Investigations) | 4 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-27): https://cdn.clinicaltrials.gov/large-docs/55/NCT01964755/Prot_SAP_000.pdf